CLINICAL TRIAL: NCT05669014
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Study of Daxdilimab Subcutaneous Injection in Adult Participants With Inadequately Controlled Dermatomyositis or Anti-synthetase Inflammatory Myositis.
Brief Title: A Phase 2 Proof of Concept Study to Evaluate the Efficacy and Safety of Daxdilimab in Participants With Dermatomyositis (DM) or Anti-synthetase Inflammatory Myositis (ASIM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZNP-DAX-205; 2022-502810-10-00 (Other: EU CT Number)
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Inflammatory Myositis
Keywords: Anti-synthetase syndrome; Myositis; Polymyositis
MeSH Terms: conditions — Myositis; Polymyositis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daxdilimab (Experimental): Daxdilimab will be administered by subcutaneous (SC) injection during the 24-week treatment period followed by an 8-week safety follow up.
  Prior to amendment 2 participants could enter an open-label extension period from weeks 24-48. For those participants already in the open-label extension, they will stop dosing and enter the safety follow up.
  Interventions: Drug: Daxdilimab
- Placebo (Placebo Comparator): Matching placebo will be administered by SC injection during the 24-week treatment period followed by an 8-week safety follow up.
  Prior to amendment 2 participants could enter an open-label extension period from weeks 24-48 and receive daxdilimab. For those participants already in the open-label extension, they will stop dosing and enter the safety follow up.
  Interventions: Drug: Daxdilimab; Drug: Placebo

INTERVENTIONS:
Drug: Daxdilimab — Participants will be administered daxdilimab by subcutaneous (SC) injection.
  Other Names: HZN-7734
Drug: Placebo — Participants will be administered identically matching placebo by SC injection.
  Arms: Placebo

SUMMARY:
The primary efficacy objective:

To evaluate the effect of daxdilimab compared with placebo in reducing disease activity at Week 24.

The secondary efficacy objectives include:

1. To evaluate the effect of daxdilimab compared with placebo in reducing disease activity at Week 24.
2. To evaluate the effect of daxdilimab compared with placebo on skin symptoms at Week 24.
3. To evaluate the effect of daxdilimab on decreasing the use of corticosteroid at Week 24.

Other secondary objectives include:

1. To characterize the pharmacokinetics (PK) and immunogenicity of daxdilimab in participants.
2. To evaluate the safety and tolerability of daxdilimab in participants.

DETAILED DESCRIPTION:
The study will enroll participants with 2 idiopathic inflammatory myositis populations:

* Population 1 or dermatomyositis (DM): participants with DM with definite or probable myositis according to the American College of Rheumatology/European League Against Rheumatism 2017 (ACR/EULAR 2017) criteria and a DM rash.
* Population 2 or anti-synthetase inflammatory myositis (ASIM): participants with ASIM with definite or probable myositis according to ACR/EULAR 2017 criteria and a positive ASIM associated antibody.

Participants will be randomized by population in a 1:1 ratio and receive investigational product (IP) daxdilimab or placebo by subcutaneous injection.

The estimated total study duration will be up to 36 weeks (up to 60 weeks for those participants who entered the open-label extension prior to amendment 2.)

Acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult men or women 18 and ≤ 75 years of age at the time of signing the informed consent (ICF).
2. A diagnosis of definite or probable myositis according to American College of Rheumatology/European League Against Rheumatism 2017 (ACR/EULAR 2017) criteria:

   1. Population 1: DM

      * Diagnosis of DM with DM rash current or historical, or
   2. Population 2: ASIM

      * Anti-histidyl tRNA synthetase-(Anti-Jo-1) antibodies must be positive during screening by central laboratory testing, or
      * One of following antibodies must be positive by historical testing: directed against anti-alanyl- (anti-PL-12), anti-threonyl-(anti PL-7), anti-asparaginyl-(anti-KS), anti-glycyl-(anti-EJ), anti-isoleucyl-(anti-OJ), anti-phenylalanyl-transfer RNA synthetase-(anti-ZO), anti-tyrosil-YRS(HA).
3. Currently active myositis with all the following (a, b, and c) during screening:

   1. Manual Muscle Testing (MMT 8) score < 142
   2. At least 2 other abnormal core set measures (CSM) from the following list:

      * Patient global disease activity (PtGDA) ≥ 2 cm in a 10 cm visual analog scale (VAS)
      * Physician's Global Disease Activity (PhGDA) ≥ 2 cm in a 10 cm VAS
      * Extramuscular activity ≥ 2cm in a 10 cm VAS
      * At least one muscle enzyme 1.5 times upper limit of normal (ULN)
      * Health assessment questionnaire-disability index (HAQ-DI) ≥ 0.5
   3. Global muscle damage score ≤ 5 on a 10 cm VAS on the myositis damage index (MDI).
4. Participants should be on stable standard of care therapy if tolerated; if they are not able to tolerate it or have failed standard of care, medications should have a washed out period.
5. Participants should be willing to taper corticosteroid dose per protocol when stable or improving.

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator or sponsor, would interfere with the evaluation of investigational product (IP) or interpretation of participant safety or study results.
2. Weight > 160 kg (352 pounds) at screening.
3. Breastfeeding or pregnant women or women who intend to become pregnant anytime from signing the ICF through 6 months after receiving the last dose of IP.
4. History of clinically meaningful cardiac disease including unstable angina, myocardial infarction, congestive heart failure within 6 months prior to randomization; arrhythmia requiring active therapy, except for clinically insignificant extra systoles, or minor conduction abnormalities; or presence of clinically meaningful abnormality on electrocardiogram (ECG) if, in the opinion of the Investigator, it would increase the risk of study participation.
5. History of cancer within the past 5 years except cutaneous basal cell or squamous cell carcinoma treated with curative therapy.
6. Any underlying condition that in the opinion of the Investigator significantly predisposes the participant to infection (eg. hepatitis C).
7. Known history of a primary immunodeficiency or an underlying condition, such as known human immunodeficiency virus (HIV) infection, or a positive result for HIV infection per central laboratory.
8. All participants will undergo testing for hepatitis B virus serology as defined in the protocol.
9. Active tuberculosis (TB), or a positive interferon gamma (IFN-γ) release assay (IGRA) test at screening, unless documented history of appropriate treatment for active or latent TB according to local guidelines.
10. Any severe herpes virus family infection (including Epstein-Barr virus, cytomegalovirus [CMV]) at any time prior to randomization.
11. Opportunistic infection requiring hospitalization or parenteral antimicrobial treatment within 2 years prior to randomization.
12. Significant organ system involvement or myositis damage (global muscle damage score > 5 on a 10 cm VAS scale on the MDI) that poses risks in the study or impedes assessments.
13. Diagnosis of immune-mediated necrotizing myopathy (IMNM) [(positive 3-hydroxy-3-methylglutaryl-coenzyme A reductase (anti-HMGR), anti-signal recognition particle (anti- SRP), or antibody negative)], inclusion body myositis (IBM) (including positive anti-cytosolic 5'-nucleotidase 1A (anti cN1A), or drug-induced myositis.
14. Current musculoskeletal, joint, or inflammatory disease, including significant joint contractures or calcinosis that in the opinion of the investigator, could interfere with the muscle strength assessments and confound the disease activity assessments.
15. Wheelchair bound participants.
16. Current inflammatory skin disease other than DM or ASIM that, in the opinion of the investigator, could interfere with the inflammatory skin assessments or confound the disease activity assessments.
17. Severe interstitial lung disease where respiratory symptoms limit participant function or progressive pulmonary fibrosis.
18. Myositis in overlap with another connective tissue disease that precludes the accurate assessment of a treatment response (for example, difficulty in assessing muscle strength in a scleroderma patient with associated myositis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of daxdilimab compared to placebo as measured by Total Improvement Score (TIS) | At Week 24
  TIS is a composite endpoint based on improvement in the 6 Disease Activity Core Set Measure (CSM) scores and range from 0 to 100 (2016 European League Against Rheumatism [EULAR]/American College of Rheumatology [ACR] Myositis Response Criteria) where a higher score is indicative of more improvement

SECONDARY OUTCOMES:
Proportion of participants with improvement of TIS ≥ 40 and without deterioration at 2 consecutive visits at 24 weeks | At 24 Weeks
  TIS is a composite endpoint based on improvement in the 6 Disease Activity Core Set Measure (CSM) scores and range from 0 to 100 (2016 European League Against Rheumatism [EULAR]/American College of Rheumatology [ACR] Myositis Response Criteria) where a higher score is indicative of more improvement
Proportion of participants with improvement of TIS ≥ 20 and without deterioration at 2 consecutive visits at 24 weeks | At 24 Weeks
  TIS is a composite endpoint based on improvement in the 6 Disease Activity Core Set Measure (CSM) scores and range from 0 to 100 (2016 European League Against Rheumatism [EULAR]/American College of Rheumatology [ACR] Myositis Response Criteria) where a higher score is indicative of more improvement
Change in the cutaneous dermatomyositis disease area and severity index (CDASI) activity score from Baseline (Day 1) to Week 24 | Baseline (Day1) to Week 24
  The CDASI is used to assess the severity of cutaneous DM and detect improvement in disease activity. The scale rates disease involvement in 15 different body areas using 3 activity (erythema, scale, erosion/ulceration) and 2 damage (poikiloderma, calcinosis) measures. The activity score ranges from 0 to 100 and the damage score from 0 to 32. Higher scores indicate greater disease severity
Proportion of participants on an oral corticosteroid (OCS) dose ≥ 10 mg of prednisone or equivalent at baseline who achieve a clinically meaningful reduction in the OCS dose at Week 24 | Baseline to Week 24
  A clinically meaningful reduction is measured as either a 25% decrease or an OCS dose of 7.5 mg/day of prednisone or equivalent
Serum concentration of daxdilimab over time | Baseline to Week 56
Proportion of the participants with anti-drug antibodies (ADA) positive post-baseline only or boosted their pre-existing ADA during the study period. | Baseline to Week 56
Incidence of ADA directed against daxdilimab over time | Baseline to Week 56
Titer of ADA to daxdilimab over time | Baseline to Week 56
Incidence of treatment emergent adverse events (TEAEs) | Baseline to Week 56
Incidence of treatment emergent serious adverse events (TESAEs) | Baseline to Week 56
Incidence of treatment emergent adverse events of special interest (TEAESIs) | Baseline to Week 56
  TEAESIs including hypersensitivity reactions, anaphylaxis, herpes zoster infection, severe [(common terminology criteria for adverse events (CTCAE)] Grade 3 or higher) viral infection/reactivation, opportunistic infection, and malignancy (except non melanoma skin cancer)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (9):
- Advanced Research Center, Inc., Anaheim, California, United States
- Brazil (2):
  - Centro Mineiro de Pesquisa - CMiP, Juiz de Fora, Minas Gerais
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
- Revmatologicky ustav, Prague, Praha, Hlavní Mesto, Czechia
- Mexico (2):
  - Unidad de Investigacion de las Enfermedades Reumaticas S.A. De C.V., Mexico City
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey
- Hospital Quironsalud Infanta Luisa, Seville, Spain
- United Kingdom (2):
  - Aintree University Hospital - NWCRN - PPDS, Liverpool, Merseyside
  - Western General Hospital Edinburgh - PPDS, Edinburgh, Midlothian

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com